CLINICAL TRIAL: NCT05593640
Title: Throboxane Effect on Chondrocytes; Role in Osteoarthritis
Brief Title: Thromboxane A2 and Osteoarthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: French Society of Rheumatology (Other)
Responsible Party: Sponsor
Other Study IDs: 22Rhumato03
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, serum and synovial liquid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ThroboxaneOA: Patient with osteoarthritis and knee effusion
  Interventions: Other: biological samples

INTERVENTIONS:
Other: biological samples — blood and synovial liquid will be sampled

SUMMARY:
TXA2 inhibits the expression of the primary marker of thermogenesis (UCP1) while prostacyclin (PGI2), another metabolite derived from arachidonic acid, enhances its expression. Given the close relationship between the adipocyte and the chondrocyte, the study team hypothesises that thromboxane A2 controls chondrocyte formation and function and thus cartilage homeostasis. The study objectives are: i) to analyse the role of TXA2 on chondrocyte differentiation in vitro, ii) to determine the association between circulating and tissue TXA2 levels in a rat model of osteoarthritis, and iii) to correlate circulating and synovial fluid levels of TXA2 with the development of osteoarthritis in a small human cohort. The proposed research aims to better understand the mechanisms underlying the role of lipid metabolites in chondrocyte formation and function, paving the way for the development of nutritional and pharmacological therapies to combat OA and associated metabolic disorders.

ELIGIBILITY:
Inclusion Criteria:

* presence of knee osteoarthritis with effusion, , no inflammatory disease

Exclusion Criteria:

* anticoagulant treatment
* inflammatory disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with osteoarthritis and knee effusion
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
to look for correlation between the rate of throboxane and the grade of osteoarthritis | 6 months
  kellgren and lawrence classification

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
not scheduled